CLINICAL TRIAL: NCT03463993
Title: Efficacy of Tranexamic Acid in Preventing Postpartum Haemorrhage After Elective Caesarean Section
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zimbabwe (Other)
Responsible Party: Principal Investigator, Chipo Gwanzura, MD, Junior Registrar, University of Zimbabwe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ETAPPPH
Record Dates: First submitted 2018-02-17; First posted 2018-03-13 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized control trial with two arms. Participants receive either 10mg/kg of TXA 10 minutes prior to elective caesarean section with prophylactic oxytocin administration after delivery of the baby, versus prophylactic oxytocin alone after delivery of the baby.
Masking Description: Trial is an open label randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Participants receive a low dose of Tranexamic acid (10mg/kg) administered slowly over 5 minutes intravenously (iv) 10 minutes prior to skin incision in elective caesarean section with prophylactic oxytocin (5 IU iv) slow administration on delivery of the baby.
  Interventions: Drug: Tranexamic Acid; Drug: Oxytocin
- Group B (Active Comparator): Participants receive prophylactic oxytocin (5 IU iv) slow administration on delivery of the baby
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Tranexamic Acid — TXA (10mg/kg) solution for injection from the vial will be diluted with 100 - 200ml electrolyte solution such as Normal Saline, Ringers solution, dextrose/water for injection on the same day it is to be used (i.e. when anaesthetist notes the patient has been randomized to receive TXA). Intravenous administration should be at a rate of 100mg or fraction thereof over at least 1 minute - usually at least 5 minutes. Standard practice is to administer over 20 minutes. Administration is to be done at least 10 minutes prior to skin incision.
  Other Names: TXA
  Arms: Group A
Drug: Oxytocin — 5IU of oxytocin are administered intravenously slowly once the baby has been delivered at caesarean section.
  Other Names: Prophylactic oxytocin

SUMMARY:
Background Postpartum haemorrhage (PPH) is a major cause of maternal mortality worldwide accounting for 25% of maternal deaths. In Zimbabwe PPH is the second most common cause of death. Tranexamic acid (TXA) is widely used to reduce blood loss in elective surgery, bleeding trauma patients, and menorrhagia.

The investigators seek to determine the efficacy of TXA in reducing PPH during and after elective caesarean section.

Methods and Design The investigators intend to perform an open label randomized control study of 1,162 women who are undergoing elective caesarean section. The participants will be randomly selected to receive an intravenous infusion of TXA 10 minutes prior to skin incision or not to receive the intervention. Prophylactic oxytocin will be administered to all the women.

The primary outcome will be incidence of PPH defined by blood loss equal to or more than 1,000ml calculated by determining the difference in haematocrit values taken prior to and 48 hours after caesarean section.

Discussion In addition to prophylactic uterotonic administration, TXA is a complementary component acting on the haemostatic process that can be used in the third stage of labour to prevent PPH. It is a promising intervention that is cheap, easy to administer and would be easy to add to routine delivery protocols in hospitals. It would also help to conserve precious resources by reducing the need for blood products, and expensive surgical interventions to manage PPH.

This large adequately powered randomized study seeks to determine the efficacy of TXA to validate its routine use at caesarean section to prevent PPH.

DETAILED DESCRIPTION:
RESEARCH QUESTION Does intravenous Tranexamic Acid (TXA) 10mg/kg plus Oxytocin 5 International Units (IU) result in a lower incidence of primary postpartum haemorrhage compared to Oxytocin alone after elective caesarean section.

RATIONALE FOR THE RESEARCH Postpartum haemorrhage (PPH) is a major cause of maternal mortality worldwide accounting for 25% of maternal deaths. In Zimbabwe, PPH is the second most common cause of death. Tranexamic acid (TXA) is widely used to reduce blood loss in elective surgery, bleeding trauma patients, and menorrhagia.

In addition to prophylactic uterotonic administration, TXA is a complementary component acting on the haemostatic process that can be used in the third stage of labour to prevent PPH. It is a promising intervention that is cheap, easy to administer and would be easy to add to routine delivery protocols in hospitals. It would also help to conserve precious resources by reducing the need for blood products, and expensive surgical interventions to manage PPH.

The investigators seek to determine the efficacy of TXA in reducing PPH during and after elective caesarean section.

RESEARCH OBJECTIVES

1. To assess the impact of TXA (10mg/kg) given 10 minutes prior to elective caesarean section on postpartum blood loss
2. To assess the potential adverse effects of TXA given 10 minutes prior to elective caesarean section Primary Outcome

   * Incidence of PPH defined by blood loss equal to or exceeding 1000ml following elective caesarean section Secondary Outcomes
   * Estimated blood loss during caesarean section
   * Need for blood transfusion
   * Use of additional uterotonics (such as oxytocin infusion or prostaglandins)
   * TXA side effects
   * Incidence of emergency surgery for PPH
   * Duration of mother's postnatal hospital stay
   * Neonatal outcome RESEARCH METHODOLOGY Research Design The aim of this study is to compare the effect of a low dose of TXA (10mg/kg) administered 10 minutes prior to elective caesarean section with prophylactic oxytocin administration, versus prophylactic oxytocin alone in an open label randomized clinical trial (RCT). An RCT is appropriate as it aims to reduce bias when testing this potentially new intervention.

Target Population Women undergoing elective caesarean sections at Harare and Parirenyatwa Hospitals based on set inclusion and exclusion criteria Inclusion criteria Pregnant woman with signed informed consent, who understand English and/or Shona, at estimated gestational age of 38 weeks or older, requiring Elective Caesarean Section, with a live intrauterine fetus.

Exclusion criteria Placental Abruption, emergency caesarean section, current or previous history of significant disease including heart disease, liver, renal disorders; known coagulopathy or history of deep venous thrombosis and/or pulmonary embolism, or arterial thrombosis (angina pectoris, myocardial infarction, stroke); history of epilepsy or seizures; autoimmune disease; sickle cell disease; severe haemorrhagic disease; intrauterine fetal demise; eclampsia/HELLP syndrome; administration of anticoagulants - clexane or antiplatelet agents in the week prior to delivery.

Sample Size A total sample size of 1,162 (581 per group) was calculated assuming a proportion of 2.1% PPH in the experimental group and 5.8% in the control group at 95% confidence interval and 90% power using Fleiss formula.

Subjects' state of physical health Healthy Intervention Participants receive either 10mg/kg of TXA 10 minutes prior to elective caesarean section with prophylactic oxytocin administration after delivery of the baby, versus prophylactic oxytocin alone after delivery of the baby.

Assessment Questionnaire (attached). Vital signs (heart rate, blood pressure, respiratory rate) noted before surgery, immediately after placental delivery, and 1 to 2 hours after birth Full blood count (FBC), Urea & electrolytes (u&e) and liver function tests (LFTs) performed a day before delivery (routinely performed) U&e, LFTs and FBC assessed 48 hours after delivery. Estimated blood loss (EBL) using the difference in hematocrit values taken prior to and 48 hours after caesarean delivery.

The investigators will also note the standard EBL based on estimates made by the anaesthetist after assessment of patient's linen and abdominal swabs.

RISKS AND BENEFITS The common adverse effects include headaches (50.4 - 60.4%), backaches (20.7 - 31.4%), nasal sinus problem (25.4%), abdominal pain (12 - 19.8%), diarrhea (12.2%), fatigue (5.2%) and anaemia (5.6%).

The WOMAN Trial collaborators found that TXA actually reduces mortality due to bleeding in women with PPH with no adverse effects.

Tranexamic acid potentiates the blood clotting system and is used to treat and prevent bleeding. Use of TXA could potentially prevent PPH due to factors other than uterine atony, where uterotonics will not be effective.

COSTS AND COMPENSATION Study participants will not receive any compensation. The cost of TXA shall not be incurred by the study participants. They will bear their usual admission and caesarean section costs that they would otherwise have borne had they not participated in the study.

INFORMED CONSENT All subjects or legally authorized representatives for minors are expected to be give informed consent.

CONFIDENTIALITY ASSURANCES Information collected from the participants shall be confidential, will be assigned a code and no personal identifiers will be used. Information collected will be stored in a secure place only accessible to the researcher and assistants, as well as on a password-protected laptop computer. Consent forms will be kept for three years after the completion of the investigation unless stipulated otherwise by the Medical Research Council of Zimbabwe.

CONFLICTS OF INTERESTS The study is being carried out in partial fulfillment of the degree of Masters of Medicine in Obstetrics and Gynaecology. No other gains are to be obtained from carrying out the study.

COLLABORATIVE AGREEMENTS N/A INTENDED USE OF RESULTS The results of the study will be submitted to the College of Health Sciences as part of the requirements for completion of the degree of Masters of Medicine in Obstetrics and Gynaecology, and may be considered for publications to add to the current body of knowledge on the use of TXA.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman with signed informed consent***
* Understand English and/or Shona
* Estimated gestational age of 38 weeks or older
* Requiring Elective Caesarean Section defined as caesarean section performed before onset of labour
* Live intrauterine fetus

  * The study will enrol participants who are Pregnant and who have a signed informed Consent form. Some of the pregnant women may be minors as they are occasionally included in patients planned for elective caesarean section for varying indications. Their inclusion also will make the results of the trial generalizable to elective caesarean section patients attended to at the two study hospitals. Consent will be sought from a legally authorized representative such as the parent or guardian.

Exclusion Criteria:

* Placental Abruption
* Emergency caesarean section
* Current or previous history of significant disease including heart disease, liver, renal disorders
* Known coagulopathy or history of deep venous thrombosis and/or pulmonary embolism, or arterial thrombosis (angina pectoris, myocardial infarction, stroke)
* History of epilepsy or seizures
* Autoimmune disease
* Sickle cell disease
* Severe haemorrhagic disease
* Intrauterine fetal demise
* Eclampsia/HELLP syndrome
* Administration of anticoagulants - clexane or antiplatelet agents in the week prior to delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2018-04-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsungai Chipato, MBChB FRCOG, Study Chair — Professor of Obstetrics and Gynaecology; Taazadza Nhemachena, MBChB MMED, Study Chair — Lecturer and Consultant; Chipo Gwanzura, MBChB, Principal Investigator — Registrar
Locations (2):
- Zimbabwe (2):
  - Harare Central Hospital, Harare
  - Parirenyatwa Group of Hospitals, Harare

IPD SHARING:
Plan to Share IPD: Yes
It is undecided whether the IPD will be made available to other researchers. Clearance is required first from ethical bodies and supervisors
Supporting Information: Study Protocol, SAP
Time Frame: TBA
Access Criteria: Communicate with researcher on chipo.gwanzura@gmail.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 8 April 2018 to 31 December 2018, we recruited 506 eligible patients. The trial was conducted at two tertiary institutions that are affiliated to the University of Zimbabwe. These serve as referral centres for 12 local authority clinics located in Harare as well as district and provincial hospitals in the surrounding provinces: Harare Central Hospital i.e. Harare Maternity Hospital (HMH) and Parirenyatwa Group of Hospitals i.e. Mbuya Nehanda Maternity Hospital (MNMH).
Period: Overall Study
Arm/Group | Group A | Group B
Started | 253 | 253
Completed | 224 | 227
Not Completed | 29 | 26
Not completed — Lost to Follow-up | 7 | 8
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 4 | 1
Not completed — Had a vaginal delivery prior to caesarean delivery | 9 | 11
Not completed — Had emergency caesarean delivery prior to elective caesarean delivery | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 224 | 227 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (6.0) | 29.7 (6.5) | 29.6 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 227 | 451
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African | 224 | 227 | 451
Region of Enrollment [Number; unit: participants]
  Zimbabwe | 224 | 227 | 451
Gestational age [Median (Inter-Quartile Range); unit: Weeks] | 39 [38 to 40] | 39 [38 to 40] | 39 [38 to 40]
HIV status [Count of Participants; unit: Participants]
  Positive | 27 | 35 | 62
  Negative | 186 | 187 | 373
  Unknown | 11 | 5 | 16
Multiple pregnancy [Count of Participants; unit: Participants] | 6 | 6 | 12
Placenta praevia [Count of Participants; unit: Participants] | 5 | 1 | 6
Uterine fibroids [Count of Participants; unit: Participants] | 5 | 1 | 6
Weight [Mean (Standard Deviation); unit: kilograms] | 78.3 (14.9) | 78.2 (15.2) | 78.3 (15.0)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.8 (5.3) | 30.5 (5.5) | 30.1 (5.4)
Number of previous caesarean sections [Count of Participants; unit: Participants]
  1 | 82 | 87 | 169
  2 | 38 | 44 | 82
  ≥3 | 5 | 13 | 18
  0 | 99 | 83 | 182
Previous surgery [Count of Participants; unit: Participants] | 10 | 11 | 21
Anaemia (Hb < 11 g/dl) [Count of Participants; unit: Participants] | 44 | 51 | 95
Foetal macrosomia (birth weight > 4000g) [Count of Participants; unit: Participants] | 8 | 6 | 14
Breech presentation [Count of Participants; unit: Participants] | 24 | 22 | 46
Risk assessment for PPH [Count of Participants; unit: Participants]
  Low | 194 | 195 | 389
  Medium | 14 | 7 | 21
  High | 16 | 25 | 41
Type of anaesthesia [Count of Participants; unit: Participants]
  General | 33 | 24 | 57
  Regional (spinal) | 176 | 188 | 364
  Missing | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postpartum Haemorrhage (PPH)
Description: PPH based on Haematocrit calculation and PPH based on Haemoglobin calculation
Time Frame: Up to 48 hours post-caesarean section
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
Participants
  PPH based on Haematocrit calculation | 48 | 54
  PPH based on Haemoglobin calculation | 56 | 71
Statistical Analysis 1: Comparison: Group A vs Group B; The null hypothesis was that intravenous Tranexamic Acid (TXA) 10mg/kg plus Oxytocin 5IU does not result in a lower incidence of primary postpartum haemorrhage compared to Oxytocin alone after elective caesarean section; Test type: Superiority; p = 0.549, Chi-squared — The p-value above is the calculated P value based on hematocrit
Statistical Analysis 2: Comparison: Group A vs Group B; The null hypothesis was that intravenous Tranexamic Acid (TXA)10mg/kg plus Oxytocin 5IU does not result in a lower incidence of primary postpartum haemorrhage compared to Oxytocin alone after elective caesarean section; Test type: Superiority; p = 0.138, Chi-squared — This is the calculated p-value based on hemoglobin

2. Secondary Outcome: Estimated Blood Loss
Description: Blood loss during caesarean section based on visual estimation and calculation.
Time Frame: At caesarean section
Population: Intention-to-treat population
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
ml
  Visually estimated blood loss | 483.73 (182.56) | 479.61 (139.49)
  Haematocrit-based calculation of estimated blood loss | 650.06 (631.50) | 653.05 (796.03)
  Haemoglobin-based calculation of estimated blood loss | 644.30 (692.27) | 707.68 (948.01)
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = 0.789, t-test, 2 sided — 0.789 is the calculated p-value for visually estimated blood loss: Visually estimated blood loss (ml): Group A mean 483.73 (standard deviation182.56); Group B 479.61 (139.49); p-value 0.789
Statistical Analysis 2: Comparison: Group A vs Group B; Test type: Superiority; p = 0.968, t-test, 2 sided — 0.968 is the calculated p-value based on hematocrit. Hematocrit-based calculation of estimated blood loss(ml): Group A mean 650.06 (standard deviation 631.50); Group B 653.05 (796.03); p-value 0.968
Statistical Analysis 3: Comparison: Group A vs Group B; Test type: Superiority; p = 0.447, t-test, 2 sided — Hemoglobin-based calculation of estimated blood loss(ml) mean(standard deviation): Group A 644.30 (692.27); Group B 707.68 (948.01); p-value 0.447

3. Secondary Outcome: Amount of Blood Transfused
Description: Requirement by participant of blood transfusion
Time Frame: At caesarean section up to 48 hours post-caesarean section
Population: Intention-to-treat population
Measure: Median (Inter-Quartile Range); unit: units of blood given
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
units of blood given | 1.5 [1 to 2] | 2.5 [2 to 3]
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Number of Participants With Use of Additional Uterotonics
Description: Number of participants who received additional uterotonics such as an oxytocin infusion or prostaglandin (misoprostol).
Time Frame: At caesarean section up to 48 hours post-caesarean section
Population: Intention-to-treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
Participants | 38 | 32
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p < 0.05, Chi-squared

5. Secondary Outcome: Number of Participants With Tranexamic Acid Side Effects
Description: Number of participants with adverse effects related to tranexamic acid use
Time Frame: From intravenous infusion of the drug up to 48 hours post-caesarean section
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
Participants | 7 | 3

6. Secondary Outcome: Number of Participants Requiring Emergency Surgery for PPH
Description: Number of participants requiring emergency surgical procedures to manage any PPH that occurs
Time Frame: At caesarean section up to 48 hours post-caesarean section
Population: Intention-to-treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
Participants | 0 | 2

7. Secondary Outcome: Number of Days of Participants' Hospital Stay
Description: The number of days the participant stayed in hospital from the date of admission to date of discharge from hospital.
Time Frame: From date of randomization until the day 2 post-caesarean section (date of discharge from hospital) or date of death whichever comes earlier
Population: Intention-to-treat population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
days | 5 [4 to 5] | 5 [4 to 5]

8. Secondary Outcome: Neonatal Outcome - Weight
Description: Neonatal birth weight in grams
Time Frame: From date of delivery of neonate by caesarean section until day 2 post-caesarean section (the date of discharge from hospital) or date of death whichever comes earlier
Population: Intention-to-treat population
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
grams | 3087.85 (523.98) | 3109.98 (513.13)

9. Secondary Outcome: Neonatal Outcome - APGAR Score of the Neonates at 1 Minute and 5 Minutes After Delivery
Description: APGAR (Appearance, Pulse, Grimace, Activity, Respiration) scores out of 10 at 1 minute and 5 minutes. A measure of the physical condition of a newborn infant. It is obtained by adding points (maximum score of 2, 1, or 0 as minimum score) for Appearance (0 - blue/pale, 1 - pink body, blue extremities, 2 - pink); Pulse (0 - absent heart rate, 1 - below 100 beats per minute, 2 - over 100 beats per minute), Grimace (Reflex irritability - 0 - floppy, 1 - minimal response to stimulation, 2- prompt response to stimulation), Activity (muscle tone: 0 - absent, 1 - Flexed arms and legs, 2 - active), Respiration ( 0 - absent, 1 - slow or irregular, 2 - vigorous cry). APGAR score at 1minute or 5 minute can be a minimum of of 0 (0+0+0+0+0) or maximum of 10 (2 for each parameter above).
Time Frame: Scores at 1 minute from time of delivery and at 5 minutes after delivery
Population: Intention-to-treat analysis
Measure: Median (Inter-Quartile Range); unit: units on a scale up to 10
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
units on a scale up to 10
  Apgar score at 1 minute | 8 [8 to 9] | 9 [8 to 9]
  Apgar score at 5 minutes | 9 [9 to 10] | 9 [9 to 10]

10. Secondary Outcome: Neonatal Outcome - Number of Neonates Admitted to the Neonatal Unit
Description: Number of neonates requiring admission to the neonatal unit from time of delivery at caesarean section
Time Frame: as for outcome 8
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
Participants | 33 | 23

11. Secondary Outcome: Neonatal Outcome - Number of Neonates Diagnosed With Jaundice
Description: Number of neonates with clinical jaundice (yellowing of the skin or whites of the eyes)
Time Frame: as for outcome 8
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
Participants | 1 | 0

12. Secondary Outcome: Neonatal Outcome - Thromboembolic Event
Description: Number of neonatal thromboembolic events
Time Frame: as for outcome 8
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
Participants | 0 | 0

13. Secondary Outcome: Neonatal Outcome - Death
Description: Neonatal death that occurs
Time Frame: as for outcome 8
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 224 | 227
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to the time the patient and baby were discharged from hospital which on average is on the third day post-caesarean section.
Description: The risk of serious adverse events is zero as these are rare events with tranexamic acid administration. The all-cause mortality is zero again as this is a rare event. The common adverse effects include headaches (50.4 - 60.4%), backaches (20.7 - 31.4%), nasal sinus congestion (25.4%), abdominal pain (12 - 19.8%), diarrhoea (12.2%), fatigue (5.2%) and anaemia (5.6%). The WOMAN Trial collaborators found that TXA reduces mortality due to bleeding in women with PPH with no adverse effects.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/224 | 0/227
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/227
Other Adverse Events (participants affected / at risk) | 7/224 | 3/227
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=224) | Group B (N=227)
Hypotension (Cardiac disorders) | 3 | 1
Headache (Nervous system disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The a priori power was not been achieved as the target sample size had not yet been achieved due to reasons beyond the scope of the study. The study had no placebo and was not blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT03463993/Prot_SAP_000.pdf